CLINICAL TRIAL: NCT00936676
Title: An Open-Label, Multi-Center, Follow-Up Study Designed to Evaluate the Long-Term Effects of Rasagiline in Parkinson's Disease Subjects Who Participated in the ADAGIO Study
Brief Title: ADAGIO Follow Up Study: Evaluation of the Long-Term Effects of Rasagiline in Parkinson's Disease Subjects
Status: Completed | Type: Observational
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Collaborators: Teva Neuroscience, Inc. (Industry); H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: TVP-1012/501; 2009-011541-24 (EudraCT Number)
Record Dates: First submitted 2009-07-08; First posted 2009-07-10 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Parkinson's Disease
Keywords: parkinson's; long-term effects; adagio; rasagiline; delayed start
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rasagiline mesylate: Enrollment by invitation to participates from the ADAGIO trial
  Interventions: Drug: rasagiline mesylate

INTERVENTIONS:
Drug: rasagiline mesylate — During the Core follow-up study period, subjects will continue to receive 1 mg rasagiline once a day. During the Extended follow-up study period, only subjects who are still on rasagiline at Visit 9 will continue to receive treatment with rasagiline 1 mg per day. Tablets will be supplied by the Sponsor and given according to the label.
  Other Names: Azilect

SUMMARY:
Eligible participants, who participated in the ADAGIO trial and who sign an approved informed consent form, will be enrolled into the study at their original study locations. participants who have stopped rasagiline therapy and in the opinion of the investigator will gain clinical benefit from restarting treatment can also be considered for enrollment in the Core follow-up study period. Use of any other anti-PD treatment is permitted as deemed necessary by the treating physician (according to the participants clinical status).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who participated in the ADAGIO study, and who entered the active phase of the study and
2. Subjects who are currently on rasagiline treatment (or subjects who have stopped rasagiline treatment, are willing to restart treatment, and in the opinion of the investigator will gain clinical benefit from restarting treatment) and
3. Subjects with a diagnosis of Parkinson's disease and
4. Subjects willing and able to give written informed consent

Exclusion Criteria:

1. Subjects who have discontinued rasagiline treatment due to an adverse event and have not restarted rasagiline treatment subsequently.
2. Subjects who cannot be given rasagiline due to any exclusion based on the local label (including pregnancy or nursing women) or due to the use of medications contraindicated for concomitant use with rasagiline according to local label
3. Subjects with a medical condition that is considered by the investigator as significant enough to prevent participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Only those who participated in the ADAGIO trial, and who sign an approved informed consent form, will be included in the follow-up study
Sampling Method: Non-Probability Sample
Enrollment: 684 (Actual)
Dates: Start 2009-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
PD Functional Status Questionnaire | 36 months
  Assess Benefits of rasagiline treatment using yes/no questions; Milestones of time to treatment-Dopaminergic treatment, levodopa, surgery for PD, time to -dyskinesia, hallucinations, functional decline using an aggregate of the responses to PD Functional Status Questionnaire
UPDRS scores | 36 months
  Part I is designed to rate mentation, behavior and mood (questions 1-4). Part II (questions 5-17) is designed to rate activities of daily life. Both parts I and II are to be collected as historical information. Part III (questions 18-31) is done as a motor examination at the time of a visit as defined in this protocol. The various items to be rated are scored using a 5-point system (i.e., 0 is normal and 4 indicates a severe abnormality, half point scores are allowed for Part III questions).
EDL scale | 36 months
Hoehn and Yahr scale | 36 months
  0 indicates asymptomatic to 5 which indicates wheelchair bound
Parkinson's Fatigue Scale | 36 months
  1 indicates strongly disagree to 5 which indicates strongly agree
Montreal Cognitive Assessment (MoCA) Scale | 36 months
  assessment of mild cognitive deficits
Non-motor symptom questionnaire of the PD Society | 36 months
  Yes/No questions
Quality of Life Questionnaire | 36 months
  Qualitative questions using Never to Always answers

CONTACTS AND LOCATIONS:
Overall Officials: C Warren Olanow, MD, FRCPC, Principal Investigator — Department of Neurology, Mount Sinai School of Medicine; Olivier Rascol, MD, Principal Investigator — Department of Clinical Pharmacology, Faculty of Medicine, University Hospital, Toulouse, France
Locations (102):
- United States (37):
  - Teva Investigational Site 7054, Birmingham, Alabama
  - Teva Investigational Site 7006, Tucson, Arizona
  - Teva Investigational Site 7018, Irvine, California
  - Teva Investigational Site 7019, La Jolla, California
  - Teva Investigational Site 7039, Loma Linda, California
  - Teva Investigational Site 7023, Los Angeles, California
  - Teva Investigational Site 7022, Sunnyvale, California
  - Teva Investigational Site 7024, Danbury, Connecticut
  - Teva Investigational Site 7016, Farmington, Connecticut
  - Teva Investigational Site 7020, Boca Raton, Florida
  - Teva Investigational Site 7011, Gainesville, Florida
  - Teva Investigational Site 7045, Miami, Florida
  - Teva Investigational Site 7017, Tampa, Florida
  - Teva Investigational Site 7055, Atlanta, Georgia
  - Teva Investigational Site 7043, Augusta, Georgia
  - Teva Investigational Site 7013, Chicago, Illinois
  - Teva Investigational Site 7052, Chicago, Illinois
  - Teva Investigational Site 7001, Northbrook, Illinois
  - Teva Investigational Site 7008, Springfield, Illinois
  - Teva Investigational Site 7037, Des Moines, Iowa
  - Teva Investigational Site 7053, Scarborough, Maine
  - Teva Investigational Site 7026, Boston, Massachusetts
  - Teva Investigational Site 7015, Lansing, Michigan
  - Teva Investigational Site 7010, Traverse City, Michigan
  - Teva Investigational Site 7029, Golden Valley, Minnesota
  - Teva Investigational Site 7004, Omaha, Nebraska
  - Teva Investigational Site 7046, Buffalo, New York
  - Teva Investigational Site 7048, Durham, North Carolina
  - Teva Investigational Site 7051, Raleigh, North Carolina
  - Teva Investigational Site 7034, Cincinnati, Ohio
  - Teva Investigational Site 7009, Toledo, Ohio
  - Teva Investigational Site 7002, Allentown, Pennsylvania
  - Teva Investigational Site 7044, Philadelphia, Pennsylvania
  - Teva Investigational Site 7050, Providence, Rhode Island
  - Teva Investigational Site 7035, Houston, Texas
  - Teva Investigational Site 7056, Houston, Texas
  - Teva Investigational Site 7025, Milwaukee, Wisconsin
- Argentina (5):
  - Teva Investigational Site 7160, Buenos Aires
  - Teva Investigational Site 7161, Buenos Aires
  - Teva Investigational Site 7162, Buenos Aires
  - Teva Investigational Site 7163, Buenos Aires
  - Teva Investigational Site 7164, Pilar - Buenos Aires
- Canada (9):
  - Teva Investigational Site 7088, Calgary, Alberta
  - Teva Investigational Site 7086, Winnipeg, Manitoba
  - Teva Investigational Site 7085, Halifax, Nova Scotia
  - Teva Investigational Site 7083, London, Ontario
  - Teva Investigational Site 7087, Markham, Ontario
  - Teva Investigational Site 7089, Toronto, Ontario
  - Teva Investigational Site 7081, Montreal, Quebec
  - Teva Investigational Site 7080, Québec, Quebec
  - Teva Investigational Site 7082, Saskatoon, Saskatchewan
- France (7):
  - Teva Investigational Site 7201, Aix-en-Provence
  - Teva Investigational Site 7202, Clermont-Ferrand
  - Teva Investigational Site 7203, Créteil
  - Teva Investigational Site 7204, Lille
  - Teva Investigational Site 7206, Nantes
  - Teva Investigational Site 7205, Pessac
  - Teva Investigational Site 7200, Toulouse
- Germany (8):
  - Teva Investigational Site 7304, Bochum
  - Teva Investigational Site 7309, Düsseldorf
  - Teva Investigational Site 7306, Erbach im Odenwald
  - Teva Investigational Site 7303, Gera
  - Teva Investigational Site 7307, Kassel
  - Teva Investigational Site 7300, Kiel
  - Teva Investigational Site 7308, Tübingen
  - Teva Investigational Site 7302, Ulm
- Hungary (3):
  - Teva Investigational Site 7400, Budapest
  - Teva Investigational Site 7401, Budapest
  - Teva Investigational Site 7404, Debrecen
- Israel (8):
  - Teva Investigational Site 7501, Ramat Gan, IL
  - Teva Investigational Site 7502, Beersheba
  - Teva Investigational Site 7504, Haifa
  - Teva Investigational Site 7507, Haifa
  - Teva Investigational Site 7505, Jerusalem
  - Teva Investigational Site 7506, Petah Tikva
  - Teva Investigational Site 7503, Ramat Gan
  - Teva Investigational Site 7500, Tel Aviv
- Italy (9):
  - Teva Investigational Site 7604, Grosseto
  - Teva Investigational Site 7600, Lido Di Camaiore (Lucca)
  - Teva Investigational Site 7602, Milan
  - Teva Investigational Site 7607, Milan
  - Teva Investigational Site 7610, Parma
  - Teva Investigational Site 7601, Pozzilli (IS)
  - Teva Investigational Site 7606, Roma
  - Teva Investigational Site 7611, Roma
  - Teva Investigational Site 7615, Roma
- Teva Investigational Site 7704, Blaricum, Netherlands
- Teva Investigational Site 7150, Lisbon, Portugal
- Romania (5):
  - Teva Investigational Site 7100, Bucharest
  - Teva Investigational Site 7102, Cluj-Napoca
  - Teva Investigational Site 7104, Constanța
  - Teva Investigational Site 7103, Târgu Mureş
  - Teva Investigational Site 7101, Timișoara
- Spain (7):
  - Teva Investigational Site 7800, Barcelona
  - Teva Investigational Site 7801, Barcelona
  - Teva Investigational Site 7802, Barcelona
  - Teva Investigational Site 7806, Bilbao
  - Teva Investigational Site 7803, Donostia / San Sebastian
  - Teva Investigational Site 7804, L'Hospitalet de Llobregat
  - Teva Investigational Site 7805, Madrid
- United Kingdom (2):
  - Teva Investigational Site 7902, Cambridge
  - Teva Investigational Site 7900, Newcastle upon Tyne

REFERENCES:
- See also: Related Info — http://clinicaltrials.gov/ct2/show/NCT00256204?term=ADAGIO&rank=1